CLINICAL TRIAL: NCT06011291
Title: A Phase I Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SYH2051 Monotherapy in Patients With Advanced Solid Tumors or in Combination With Radiotherapy in Patients With Locally Advanced Head and Neck Cancer
Brief Title: A Study of SYH2051 Monotherapy in Advanced Solid Tumors or in Combination With Radiotherapy in Locally Advanced Head and Neck Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYH2051-001
Record Dates: First submitted 2023-08-14; First posted 2023-08-25 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Solid Tumors; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: SYH2051 monotherapy dose escalation in advanced solid tumors (Phase Ia) (Experimental)
  Interventions: Drug: SYH2051 tablets
- Arm B: SYH2051+RT dose escalation in locally advanced head and neck cancer (Phase Ib) (Experimental)
  Interventions: Drug: SYH2051 tablets; Radiation: Intensity-Modulated Radiation Therapy (IMRT)
- Arm C: SYH2051+RT dose expansion in locally advanced head and neck cancer (Phase Ic) (Experimental)
  Interventions: Drug: SYH2051 tablets; Radiation: Intensity-Modulated Radiation Therapy (IMRT)

INTERVENTIONS:
Drug: SYH2051 tablets — Arm A: Five dose levels will be administered sequentially. Arm B and C: Concurrently administered with RT, and 2 weeks adjuvant treatment after RT.
Radiation: Intensity-Modulated Radiation Therapy (IMRT) — Radical or adjuvant radiotherapy
  Arms: Arm B: SYH2051+RT dose escalation in locally advanced head and neck cancer (Phase Ib); Arm C: SYH2051+RT dose expansion in locally advanced head and neck cancer (Phase Ic)

SUMMARY:
This is an open-label, multicenter, dose-escalation phase I study to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor efficacy of SYH2051 in patients with advanced solid tumors or in combination with radiotherapy (RT) in patients with locally advanced head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. Phase Ia: Patients with histologically or cytologically confirmed advanced solid tumors, for whom there is no standard therapy available, or ineffective or intolerant to standard therapy. Phase Ib/Ic: Patients with histologically or cytologically confirmed locally advanced head and neck cancer suitable for radiotherapy alone;
3. Eastern Collaborative Oncology Group (ECOG) Performance Status of 0~1;
4. Patients in medical conditions to be able to receive radiotherapy (for phase Ib/Ic);
5. Life expectancy of >3 months;
6. At least one measurable lesion (excluding patients in phase Ic combined with adjuvant radiotherapy);
7. Patients with adequate hematologic, hepatic, renal and coagulation function;
8. Patients are not pregnant or lactating and required contraception;
9. Patients who are willing to provide written informed consent form (ICF) before the beginning of the study.

Exclusion Criteria:

1. Any antineoplastic therapy such as chemotherapy, biologic therapy, endocrine therapy, or immunotherapy within 4 weeks before the first dose of the study drug (or within 5 half-lives of other unmarketed study drugs, whichever is longer), except for the following:

   1. 6 weeks for Nitrosoureas or mitomycin C;
   2. 2 weeks or five half-lives (whichever is longer) for oral fluorouracil and small molecule targeted drugs;
   3. 2 weeks for Chinese herbal medicine with antineoplastic indications;
2. Patients with previous (within 2 years before screening) or concurrent other malignancies (only for phase Ib/Ic);
3. Patients had undergone major organ surgery (excluding needle biopsies) within 4 weeks before the first dose, with obvious trauma, or require elective surgery during the study;
4. Severe, non-healing fractures within 4 weeks before the first dose of the study drug;
5. The adverse reactions of previous antineoplastic therapy have not recovered to ≤grade 1 as determined by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria;
6. Patients who had received treatment with any drug that is a medium or strong inhibitor or inducer of cytochrome P450 (CYP) 3A4/5 enzyme activity within 2 weeks before screening or need to continue receiving such drugs;
7. Active brain metastases and/or carcinomatous meningitis;
8. Concurrent serious and/or uncontrolled medical conditions at screening (e.g., severe chronic obstructive pulmonary disease);
9. Patients with abnormal thyroid function were not allowed, except those with euthyroid function after drug control;
10. History of severe cardiovascular disease;
11. History of myopathy or raised creatine kinase (CK) >5 times the upper limit of normal (ULN);
12. Known hypersensitivity or intolerance to any component of the study drug or its excipients;
13. History of autoimmune disease, immunodeficiency disease, including HIV testing positive or other acquired, congenital immunodeficiency diseases, or organ transplantation;
14. Active hepatitis B virus, hepatitis C virus or active syphilis infection;
15. Active dysphagia, malabsorption or other chronic gastrointestinal diseases or conditions that may hamper compliance and/or absorption of the study drug;
16. Other ineligibilities according to the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | 31 days for Arm A and 11 weeks for Arm B
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 2 years
Maximum tolerated dose (MTD)(if any) or maximum administrated dose (MAD) | up to 1 year
Recommended phase 2 dose (RP2D) of SYH2051 in combination with RT | 2 years

SECONDARY OUTCOMES:
Phase Ia: Maximum Plasma Concentration (Cmax) | 1 years
Phase Ia: Time to Maximum Plasma Concentration (Tmax) | 1 years
Phase Ia: Area under the plasma concentration-time curve from time zero to time of last measurable concentration(AUC0-last) | 1 years
Phase Ia: Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) | 1 years
Objective response rate (ORR) | 2 years
Disease Control Rate (DCR) | 2 years
Duration of locoregional control (DoLC) | 2 years
Phase Ib and Ic: Concentrations of SYH2051 | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Information Group, Shijiazhuang, Hebei, China